CLINICAL TRIAL: NCT01860716
Title: Impact of Melatonin in the Pretreatment of Organ Donor and the Influence in the Evolution of Liver Transplant: a Prospective, Randomised Double-blind Study.
Brief Title: Impact of Melatonin in the Pretreatment of Organ Donor and the Influence in the Evolution of Liver Transplant.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aragon Institute of Health Sciences (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PI10/02877
Record Dates: First submitted 2013-05-17; First posted 2013-05-23 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Evidence of Liver Transplantation
Keywords: Melatonin, liver transplant, oxidative stress
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Solution for infusion (Placebo Comparator): Solution for infusion administrated via nasogastric tube
  Interventions: Drug: Placebo
- Melatonin (Experimental): 30 mg melatonin administrated via nasogastric tube in the Intensive Care Unit when included in the study and 30 mg melatonin 60 minutes before transfer to the operating room.
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — Melatonin 2 mg prolonged-release tablet, administration via nasogastric tube.
  Other Names: Circadin (Neurim Pharmaceuticals)
  Arms: Melatonin
Drug: Placebo
  Arms: Solution for infusion

SUMMARY:
Impact of melatonin on organ donor pretreatment and liver transplant recipient: prospective, randomized, double-blind trial.

OBJECTIVES. To establish the efficacy of the melatonin administered to encephalic death donors (EDD) in liver transplantation. The aim is to improve the functional quality of the retrieved organs, attenuate lesions and ischemia-reperfusion mediators, and provide grafts with greater resistance to post-transplant aggression.

METHODOLOGY. Prospective, randomized, double-blind, pilot trial to evaluate preconditioning with melatonin versus placebo in EDDs. Two groups, melatonin and control-placebo, n=30 per group. Administration to donor via NG tube of 30mg of melatonin or placebo (lactose) upon inclusion in the trial, 60 minutes prior to commencement of surgery and following laparotomy during extraction. Evaluation of response to treatment: A) Conventional clinical, hemodynamic, analytical and histopathological parameters in donor and recipient. B) Plasma determinations for: oxidative/nitrosative stress; acute phase proteins; cellular and humoral immunity; NT-proBNP and cystatin C; endocrine profile; melatonin levels. C) Determinations in liver tissue: quantification of malonyldialdehyde-4hydroxyalkenals and protein carbonyl content; cellular and mitochondrial membrane fluidity; markers of tissue-vascular damage and proliferation: transforming growth factor-beta (TGF-β); hypoxia-inducible factor (HIF) and vascular endothelial growth factor (VEGF). Data will be analyzed following a prospectively define plan and by intention-to-treat analysis.

DETAILED DESCRIPTION:
This study will be done in the Hospital Clinico Lozano Blesa (Zaragoza, Spain), promoted by the Health Science Aragon Institute and its principal investigator is F. Agustín García Gil (Surgical Service). It will start in April-May 2013 and will finish 12 months later approximately. The study sponsor is I+CS (Aragon Institute of Health Sciences).

ELIGIBILITY:
Inclusion Criteria:

A) Donors

1. Encephalic-death (ED) organ donor who is situated in the ICUs of accredited hospitals in Zaragoza and meets each and every one of the following criteria.
2. Being 16 years old or older.
3. Informed consent for the donation signed by the immediate family.
4. Informed consent for inclusion of the donor in the study .
5. Receive intensive treatment and standard maintenance of the donor in ED, in accordance with universally accepted protocols of the Organizacion Nacional de Trasplantes (ONT), of the Aragon Autonomous Transplant Coordination, and of the ICUs and the participating hospitals in the study.

B) Liver transplant recipients

1. Being 18 years old or older and being less than 68 years of age.
2. Informed consent for the procedure of LT signed.
3. Informed consent for patient inclusion in the study, signed the same day that consent to the LT.

Exclusion Criteria:

A) Donors

A potential encephalic-death organ donor will not be included in the study if either of the following criteria:

1. Absence of either signed informed consent: for organ donation or for inclusion in the study.
2. No standard concomitant treatment and management of donor in ED.

B) Liver transplant recipients

1. Absence of either signed informed consent: for liver transplantation or for inclusion in the study.
2. Split, domino or multiorgan transplantation.
3. Grafts removed by other surgical teams.
4. Pregnant women or fertile not using contraceptive measures highly effective.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
AST levels | Between days 1 and 10 postoperatively.
  Aspartate transaminase (AST) levels will be measured.
ALT | Between days 1 and 10 postoperatively
  Alanine transaminase (ALT) levels will be measured.
Bilirubin levels | Between days 1 and 10 postoperatively
  Bilirubin levels will be measured.
Prothrombin levels | Between days 1 and 10 postoperatively
  Prothrombin levels will be measured.

SECONDARY OUTCOMES:
Post-reperfusion syndrome | Transplant day
  Post-reperfusion syndrome
No primary function and primary graft dysfunction | Transplant day
  No primary function and primary graft dysfunction
Survival of the graft | From day 0 to 3 months
  Survival of the graft
Patient survival | Day 0 to 3 months
  Patient survival
Donor and recipient serological parameters | Between days 1 and 10 postoperatively
  Donor and recipient serological parameters
Morphological and functional quality of the liver graft evaluated by histological parameters of ischemia-reperfusion and tissue biochemical markers | Day 0 and day 1
  Morphological and functional quality of the liver graft evaluated by histological parameters of ischemia-reperfusion and tissue biochemical markers

CONTACTS AND LOCATIONS:
Overall Officials: Francisco A. García-Gil, Physician, Principal Investigator — Hospital Clínico Universitario Lozano Blesa
Locations (1):
- Hospital Clínico Universitario Lozano Blesa, Zaragoza, Zaragoza, Spain